CLINICAL TRIAL: NCT05317130
Title: A Complex Health Promotion Intervention in Parasport - The Safe & Healthy Parasport Project
Status: Not yet recruiting | Type: Observational
Sponsor: Lund University (Other)
Collaborators: University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Kristina Fagher, Principal Investigator, Lund University
Other Study IDs: Safeparasport
Record Dates: First submitted 2022-02-14; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Sport Injury; Diabetes; Health Behavior; Illness Behavior; Literacy
Keywords: Para sport; Sports injuries; Athlete health; Health promotion; Health literacy
MeSH Terms: conditions — Diabetes Mellitus; Health Behavior; Illness Behavior; Literacy; Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- This is an observational study.: The cohort will consist of elite Para athletes (athletes with an impairment).
  Interventions: Other: Athlete health monitoring

INTERVENTIONS:
Other: Athlete health monitoring — Observational study

SUMMARY:
The interest in Para sport is steadily increasing. A concern is, though, that elite Para athletes report a high incidence of injuries and illnesses. Altogether, there is an urgent need to prevent such incidents among athletes already suffering from an impairment. However, most of the existing training-based prevention programmes are not adapted or accessible to Para athletes. Also, recent research suggests that sports safety work advantageously should facilitate disease prevention and health promotion. Such intervention would hypothetically also have the potential to reduce injuries, illnesses and improve health among Para athletes. To allow full implementation, the intervention would need to be adapted to the Para athletes´ various impairments, abilities and sports.

MAIN QUESTIONS TO BE ADRESSED

* Can an evidence-based eHealth health promotion platform prevent sports injuries and illnesses in elite para athletes over 6 months, 12 months and 5 years?
* Can such platform improve overall health parameters such as sleep, nutrition and mental health in elite para athletes and influence the performance parameters training quantity and training quality over 6 months, 12 months and 5 years?
* Can such platform improve health literacy among Para athletes?

DETAILED DESCRIPTION:
Introduction Sport is today one of the largest movements in Sweden, with more than three million people being members of a sports club. Participation in sport leads to several health benefits as it improves both physical and mental health. For example, it reduces the risk for cardiometabolic disease, fractures, dementia, mental illness and some cancer types. Sport also supports the development of social skills during different periods in people's lifetime. Sport has therefore a great impact on the quality of life for the individual person as well as for our health economics, as it can prevent and treat disease. The interest in sport and its associated benefits for persons with an impairment (Para sport) has also increased in the last few decades. Para sport is, however, still a young sporting discipline and despite the fact that sport poses the athlete at a risk for suffering a sports-related injury or illness few studies have assessed the burden of such incidents in Para sport.

The Para athlete and Paralympic athlete What characterises Para and Paralympic athletes is the existing impairment, whether it is physical, visual or intellectual. According to the World Health Organization the definition of an impairment is: "a problem in body function or structure" (WHO). Depending on the nature of the impairment the athlete may also have a greater risk for suffering from secondary health complaints, early age related health conditions, health risk behaviours and higher rates of premature death.

For example, individuals with SCI may be predisposed to infections, skin breakdown, osteoporosis, contractures, spasticity, pain, depression, fatigue, hyperthermia, bowel dysfunction and cardiorespiratory insufficiency. Several of these health complaints may also be present in individuals with other neurological diseases such as multiple sclerosis (MS), stroke, traumatic brain injury and cerebral palsy (CP). Individuals with more rare diagnosis such as Becker muscular dystrophy, Duchenne muscular dystrophy and Friedreich's ataxia may in addition suffer from health complaints such as heart arrhythmias and a malformed skeleton. Joint contractures and muscle fibrosis are present in individuals with arthrogryposis, which often leads to musculoskeletal problems. The biomechanics is often altered among individuals with limb deficiency, which may cause stress fractures, tendinopathies and osteoarthritis. Also stump conditions such as phantom pain, rashes and heterotopic ossification are common. Furthermore, alterations in the vascular physiology may induce cardiac disease.

Individuals with visual impairment have in general a greater risk for morbidity and unintentional injury and illness such as cardiometabolic disease, depression, falls and fractures. Other health conditions that are sometimes present with diagnoses related to visual impairments are joint problems, obesity, hearing impairment, diabetes and development delay. Individuals with intellectual impairments have more often a poor mental and physical health compared to the rest of population. Higher rates of health complaints, such as gastrointestinal disease, obesity, epilepsy, cardiometabolic disease and mental illness have been reported. Altogether, the Para athlete has other conditions due to the impairment and the sometimes associated health complaints when entering sports in comparison with an able-bodied athlete, which possibly could affect training behaviour as well as the epidemiology and consequences of sports-related injuries and illnesses.

Epidemiology of sports-related injuries and illnesses Despite all the positive health effects of sports, sports-related injuries and illnesses are a concern in most elite sports settings, as they may lead to morbidity, an ending of the sport career, long- term disability and mortality. Sports-related injuries are also a cost and burden for society.

Traumatic sports injuries, such as concussion, ligament sprains, joint distortions or fractures may, for example, lead to brain damage, osteoarthritis and chronic pain for the individual athlete. Catastrophic injuries leading to spinal injuries and death are less common, but still a concern in several sports. Overuse-related injuries may also cause several health complaints such as inflammation, degeneration and chronic pain. Recent research has suggested that the risks associated with sports- related injuries and its consequences are unacceptable when evaluated against acceptable criteria from occupational health.

Sports-related illnesses have also received more focus during the last decade. However, studies concerning the epidemiology of sports-related illnesses are still underrepresented in comparison to sports injury epidemiology. A concern is that there still are few cohort studies concerning sports injury and illness epidemiology in Para sport. Moreover, definitions and data collection methods have not been adapted to the Para athletes´ various impairments. To assist the development of evidence-based preventive measures the aim of my PhD-thesis was to gain an in-depth understanding of the epidemiology and data collection methods of sports injuries and illnesses in Para athletes. First an eHealth application for self-reported data collection of injuries and illnesses adapted to the Web Content Accessibility guidelines and Para athletes was developed and evaluated in a pilot feasibility and usability study. Thereafter, 107 Swedish elite para athletes were followed prospectively during 52 weeks. In the thesis, which is the first study globally that prospectively has followed a large cohort of Para athletes, it was shown that 68% reported an injury and 77% an illness, which is a higher incidence compared to able-bodied athletes in Sweden. One third of the injuries were classified as severe and the athletes´ impairment was involved in the mechanism in 59% of the injuries. For example, wheelchair athletes reported a high proportion of shoulder injuries and athletes with VI reported falls. Also diagnoses such as spasticity and neurogenic bladder were reported, which are not seen in able-bodied athletes. Two thirds of the athletes reported poor sleep, 48% reported persistent pain and 34% reported anxiety. Data also show that more injuries are reported at the Paralympic Games compared to the Olympic Games. Altogether, there is an urgent need to further understand the epidemiology of sports injuries and illnesses, and to prevent injuries and illnesses in Para athletes.

A concern is that the development and evaluation of evidence-based prevention strategies take time. However, research among able-bodied athletes has shown that regular athlete health monitoring with accompanied medical guidance may reduce the burden of sports injuries and illnesses, and shorten the time loss from sport when injured/ill. The medical team following up the athlete should consist of qualified and experienced individuals operating in synergy with the coach and the athlete towards a common performance and health goal. It has been proposed that this system facilitate a balanced approach to training and competing decisions, especially while the athlete is ill or injured. This method can be supported by results from my PhD-thesis, in which it it was shown that 90% of the athletes found it important to conduct athlete health monitoring also in the future. Moreover, qualitative data have revealed that Para athletes´ perceptions are that they do not have the same prerequisites as able-bodied athletes when being injured or ill. In summary, it can be hypothesized that regular athlete health monitoring over time will help us to further improve our understanding of the epidemiology of sports injuries and illnesses in Parasport, and that immediate medical guidance also can minimize the impact of a sports injury or illness.

Health promotion in sports Another concern in Parasport is that the existing prevention programmes in sports such as the knee control are not adapted to Para athletes, as several athletes are wheelchair users or amputees. Among able-bodied athletes, it has been recommended that sports safety work should facilitate health promotion, including health education. A recent study of able-bodied Swedish athletes have shown that a health promotion webpage for elite athletics athletes can reduce the injury risk. However, there is no health promotion webpage for Swedish Para athletes.

Taken together an accessible eHealh based health promotion platform will first be developed in this project using a participatory action based research design. Thereafter the following research questions will be adressed:

* Can an evidence-based eHealth health promotion platform prevent sports injuries and illnesses in elite para athletes over 6 months, 12 months and 5 years?
* Can such platform improve overall health parameters such as sleep, nutrition and mental health in elite para athletes and influence the performance parameters training quantity and training quality over 6 months, 12 months and 5 years?
* Can such platform improve health literacy among Para athletes?

ELIGIBILITY:
Inclusion Criteria:

* Being an registered para athlete in Sweden or South Africa
* Having an athlete classification according to the International Paralympic Committee

Exclusion Criteria:

* Age below 18 years, or older than 66
* Being a non-classified athlete

Ages: 18 Years to 66 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants from the Swedish and South African Paralympic programmes will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of sports injuries and illnesses 6 months following study start | The incidence will be followed up 6 months following study start
  The incidence of sports injuries and illnesses is the primary outcome. Incidence data will be calculated as the number of injuries and illnesses per 1000 hours of sports exposure.
Incidence of sports injuries and illnesses 12 months following study start | The incidence will be followed up 12 months following study start
  The incidence of sports injuries and illnesses is the primary outcome. Incidence data will be calculated as the number of injuries and illnesses per 1000 hours of sports exposure.
Incidence of sports injuries and illnesses 4 years following study start | The incidence will be followed up 4 years following study start
  The incidence of sports injuries and illnesses is the primary outcome. Incidence data will be calculated as the number of injuries and illnesses per 1000 hours of sports exposure.

SECONDARY OUTCOMES:
Mental health 6 months following study start. | Athlete mental health data will be followed up 6 months following study start.
  A secondary outcome is mental health (anxiety and depressing using the PHQ4-questionniare)
Mental health 12 months following study start. | Athlete mental health data will be followed up 12 months following study start.
  A secondary outcome is mental health (anxiety and depressing using the PHQ4-questionniare)
Mental health 4 years following study start. | Athlete mental health data will be followed up 4 years following study start.
  A secondary outcome is mental health (anxiety and depressing using the PHQ4-questionniare)
Health literacy 6 months following study start. | Health literacy data will be followed up 6 months following study start.
  A secondary outcome is health literacy (using theThe European Health Literacy Survey Questionnaire (HLS-EU-Q47)
Health literacy 12 months following study start. | Health literacy data will be followed up 12 months following study start.
  A secondary outcome is health literacy (using theThe European Health Literacy Survey Questionnaire (HLS-EU-Q47)

CONTACTS AND LOCATIONS:
Locations (1):
- Lund University, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No
The is no plan to share IPD data with other researchers.